CLINICAL TRIAL: NCT03006146
Title: Evaluation of a Single Dose of Inhaled Sargramostim in Patients With Autoimmune Pulmonary Alveolar Proteinosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Rare Diseases Clinical Research Network (Network); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TPSC-110; UL1TR001425 (NIH)
Record Dates: First submitted 2016-11-28; First posted 2016-12-30 (Estimated); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Autoimmune Pulmonary Alveolar Proteinosis
MeSH Terms: conditions — Pulmonary Alveolar Proteinosis, Acquired | interventions — sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sargramostim (Experimental): Participants will receive a single administration of inhaled sargramostim (either 125 mcg or 250 mcg dose)
  Interventions: Drug: Sargramostim

INTERVENTIONS:
Drug: Sargramostim — Participants will receive a single administration of inhaled sargramostim (either 125 mcg or 250 mcg dose)
  Other Names: Leukine; recombinant human GM-CSF

SUMMARY:
Autoimmune PAP is a rare lung disease affecting less than 5,000 individuals in US with no FDA-approved pharmacologic therapy. Results from "off-label" use in case reports and clinical studies completed outside of the US indicate that inhaled rhGM-CSF may be a safe and effective thera-py for autoimmune PAP. Preliminary clinical trials of inhaled rhGM-CSF in autoimmune PAP patients show promising results, 62%-96% therapeutic response rate without any identifiable drug-related adverse effects in at least 73 autoimmune PAP patients. However, the pharmacokinetics (PK), pharmacodynamics (PD), optimal dose, and treatment duration to maximize efficacy are unknown.

The goal is to begin to address these knowledge gaps for inhaled sargramostim for autoimmune PAP patients with a pilot safety and PK/PD study (TPSC-110). TPSC-110, PharmPAP, which is a self-controlled open-label, phase I study to evaluate the safety, PK, and PD of inhaled sargra-mostim in autoimmune PAP patients. These results will impact the field by 1) confirming existing published data, 2) monitoring the local effects of inhaled sargramostim in autoimmune PAP patients, 3) potentially demonstrating a safe starting dose for a later trial to evaluate the therapeutic efficacy of inhaled sargramostim for autoimmune PAP.

DETAILED DESCRIPTION:
PAP is a rare syndrome of surfactant accumulation and resulting hypoxemic respiratory failure that occurs in a number of diseases classified pathogenically into three groups: primary PAP (caused by disruption of GM-CSF signaling - autoimmune PAP, hereditary PAP), secondary PAP (caused by reduction in alveolar macrophage numbers and/or functions), and surfactant dysfunction-related PAP (caused by mutations in genes required for normal surfactant production). In current clinical practice, PAP is diagnosed based on a lung biopsy; an approach that is not able to identify the etiology of the PAP. Current therapy involves the physical removal of surfactant by a procedure in which the lungs are repeatedly filled with saline and emptied - whole lung lavage, which is invasive, inefficient, and not widely available, especially for children. Importantly, research advances have elucidated the pathogenesis of diseases causing PAP in most patients and have identified new diagnostic and therapeutic approaches. Simple blood-based research tests can now identify the PAP-causing disease in about 95% of patients. Further, several promising potential disease-specific therapies are currently in development. Preliminary clinical trials of inhaled rhGM-CSF in autoimmune PAP patients show promising results, 62%-96% therapeutic response rate at two doses (250 and 500 mcg/day) without any identified safety concerns. At least 73 people with autoimmune PAP have been reported to have received inhaled sargramostim with no identified drug-related adverse effects. However, the PK, PD, optimal dose, and treatment duration needed to maximize efficacy are unknown. The short-term goal is to address knowledge gaps for inhaled sargramostim for autoimmune PAP patients in the following clinical study: a pilot safety and PK/PD study (TPSC-110). A major goal of this protocol is to evaluate the local and systemic safety, PK, and PD one dose of inhaled sargramostim in autoimmune PAP. The central hypothesis is that in patients with autoimmune PAP, aerosol inhalation of sargramostim will be well-tolerated and safe because the GM-CSF autoantibody will limit detection of free GM-CSF thereby preventing local and systemic toxicity. The specific objectives of this study are to: 1) evaluate the safety profile of one dose of inhaled sargramostim in patients with autoimmune PAP 2) estimate the PK profile of inhaled sargramostim following single dose administration in patients with autoimmune PAP 3) measure the PD effects of inhaled sargramostim following single dose administration in patients with autoimmune PAP.

The target population is adults with autoimmune PAP who have measurable, clinically significant disease satisfying all of the inclusion and exclusion criteria. The study design will involve recruitment, screening, and enrollment of participants into a phase I, open-label, multi-site study. Sargramostim will be administered to autoimmune PAP patients via aerosol inhalation one time at a dose of 125 mcg or 250 mcg. Adverse events (AEs), serious AEs (SAEs), PK, and PD parameters will be evaluated (see Appendix 3 Schedule of Events). The experimental approach will evaluate 1) safety of inhaled sargramostim by documenting occurrence of treatment-emergent AEs and SAEs, 2) PK profile of GM-CSF in serum and BAL fluid, 3) local and systemic PD effects of inhaled GM-CSF and 4) effects of inhaled GM-CSF on the quality of life for participants. Anticipated results will determine the safety profile of inhaled sargramostim in patients with autoimmune PAP, will evaluate total and free GM-CSF levels in blood and lung, effects of sargramostim on blood and BAL cell counts, differentials, baseline- and GM-CSF-responsiveness of blood leukocytes and BAL cells, and biomarkers of PAP in patients with autoimmune PAP after single dose administration. These results will impact the field by 1) confirming existing published data, 2) monitoring local effects of inhaled sargramostim in autoimmune PAP patients, 3) demonstrating a safe starting dose to evaluate the efficacy of inhaled sargramostim for autoimmune PAP.

ELIGIBILITY:
Inclusion Criteria:

Male or female

Age ≥ 18 years and ≤ 80 years

Able to understand and willing to sign a written informed consent document

Able and willing to use hand held nebulizer

Able and willing to adhere to study visit schedule and study procedures

Diagnosis of autoimmune PAP determined by:

* History of a diagnosis of PAP with or without supporting lung histology or BAL/cytology

and

* Abnormal serum GM-CSF autoantibody test (GMAb ELISA Test)

and

* Chest CT findings compatible with a diagnosis of autoimmune PAP

Evidence of impaired GM-CSF signaling demonstrated by an abnormal STAT5 phosphorylation index (STAT5-PI) test measured in heparinized whole blood at the time screening

A-aDO2 ≥ 15 mm Hg

Exclusion Criteria:

Diagnosis of any other PAP-causing disease

Autoimmune PAP complicated by:

* Severe disease at screening/enrollment (A-aD02<50)
* Clinically significant pulmonary fibrosis

History of any clinically significant:

* Other lung disease
* Cardiovascular disease
* Disease requiring use of systemic steroids in past year
* Coagulopathy or other hematologic disease
* Active / serious lung or systemic infection
* Persistent or unexplained fever >101oF within 2 months of study
* Use of any immunosuppressive medication within 3-6 months of screening
* Women who are pregnant or plan to become pregnant
* History of active tobacco/e-cig/marijuana use
* Concomitant or recent use of specific medicines

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-07-13 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2021-06-07 (Actual)

PRIMARY OUTCOMES:
Occurrence of any treatment-emergent adverse events and serious adverse events | 1 year
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Maximum plasma GM-CSF Concentration (Cmax) | 1 year
  Maximum concentration of free and toal GM-CSF in the plasma following a single administration of inhaled sargramostim
Time to maximum plasma GM-CSF concentration (TMax) | 1 year
  Time to maximum plasma concentrations of free and total GM-CSF following a single administration of inhaled sargramostim
GM-CSF Area Under the Curve (AUC) | 1 year
  Systemic exposure to GM-CSF in plasma samples collected at regular intervals following a single administration of inhaled sargramostim
Half-life of inhaled GM-CSF (t1/2) | 1 year
  Half-life of GM-CSF following a single administration of inhaled sargramostim
Complete cell counts and differentials in blood and BAL fluid | 1 year
  Cell Counts and differentials in blood and BAL fluid following a single administration of inhaled sargramostim will be compared to baseline values (pre-study drug administration)
GM-CSF autoantibody levels in blood and BAL fluid | 1 year
  GM-CSF autoantibody concentrations in blood and BAL fluid following a single administration of inhaled sargramostim will be compared to baseline values (pre-study drug administration)
GM-CSF signaling levels in blood and BAL fluid | 1 year
  Responsiveness of blood and BAL cells to in vitro stimulation with GM-CSF in blood and BAL fluid following a single administration of inhaled sargramostim will be compared to baseline values (pre-study drug administration)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Trapnell, Study Chair — Children's Hospital Medical Center, Cincinnati
Locations (2):
- United States (2):
  - University of California, Los Angeles, Los Altos, California
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No